CLINICAL TRIAL: NCT02444390
Title: Identification of the Molecular Alterations Associated With Resistance to Endocrine Therapy and Impacting Treatment With mTOR Inhibitor of HR+ Metastatic Breast Cancer in Post-menopausal Women
Brief Title: Molecular Alterations Associated With Resistance to Endocrine Therapy and Impacting Treatment With mTOR Inhibitor
Acronym: SAFIR-TOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Novartis (Industry); Fondation ARC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UC-0105/1403
Record Dates: First submitted 2015-05-11; First posted 2015-05-14 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Breast Cancer
Keywords: Failed non steroidal aromatases inhibitors; Eligible for everolimus+exemestane
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exemestane+everolimus (Other): Exemestane+everolimus are administered as per their approved indication
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — biopsy of a metastasis

SUMMARY:
This is a prospective biomarker study to show that p4EBP1 staining predicts clinical benefit from treatment with everolimus in patients who are eligible for everolimus+exemestane treatment. This trial is not aimed at evaluating a drug activity. Everolimus and exemestane are prescribed within their approved indication as per usual practice and are not part of this trial.

DETAILED DESCRIPTION:
Estrogen hormone receptor-positive metastatic breast cancer who failed to non steroidal aromatases inhibitors in patients who are eligible for everolimus+exemestane treatment

ELIGIBILITY:
Inclusion Criteria:

- Eligible for everolimus+exemestane treatment as required by the marketing authorisation conditions

1. Women (or men) with histologically-proven Estrogen Receptor-positive (ER+) and/or Progesterone Receptor-positive (PR+) / Human Epidermal growth factor Receptor 2-negative (HER2-) metastatic breast adenocarcinoma or locally advanced disease who cannot be treated with surgery and/or radiation therapy
2. Postmenopausal women
3. Asymptomatic if visceral disease
4. Second line hormonotherapy or more for metastatic or locally advanced disease after recurrence or progression following a non-steroidal aromatase inhibitor (in adjuvant or metastatic setting)

   - Eligible for the biopsy
5. Progressive disease under endocrine therapy at the time of inclusion
6. Treatment with everolimus and exemestane not yet started
7. Patients with metastases that can be biopsied, except bone metastases
8. Measurable or evaluable disease
9. Age ≥18 years
10. WHO Performance Status 0/1
11. Provision of signed and dated, written informed consent prior to any protocol specific procedure, including biopsy
12. Patient with social insurance coverage

Exclusion Criteria:

1. Contraindications for everolimus+exemestane treatment
2. Previous treatment with an anti-mTOR therapy
3. More than 1 previous line of chemotherapy in metastatic setting
4. Life expectancy <3 months
5. Spinal cord compression and/or symptomatic or progressive brain metastases (unless asymptomatic or treated and stable off steroids for at least 30 days prior to start of study drug)
6. Haematopoietic function or organ impairment as shown by the following criteria:

   * Polynuclear neutrophils <1.5 x 10⁹/L
   * Platelets <100 x 10⁹/L
   * Haemoglobin <90 g/L
   * Alanine aminotransferase (ALAT) / aspartate aminotransferase (ASAT) >2.5 x ULN in the absence of or >5 x upper limit of normal (ULN) in the presence of liver metastases
   * Bilirubin >1.5 x ULN
   * Creatinine clearance ≤50 mL/min (measured or calculated by Cockcroft and Gault formula)
   * Calcium and phosphate >ULN
7. Abnormal coagulation or any other medical situation contraindicating biopsy
8. Bone metastases when this is the only site of biopsiable disease
9. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol
10. Individuals deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-05-19 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
the predictive value of p4EBP1 for an mTOR inhibitor efficacy | from inclusion up to 6 months
  The primary endpoint of the trial is the predictive value of p4EBP1 for an mTOR inhibitor efficacy, measured by the association between expression level of the biomarker (high vs low expression with a cutoff value set at the median percentages of marked cells) and clinical benefit after 6 months of everolimus+exemestane treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bachelot, MD, Principal Investigator — Centre Léon Bérard, Lyon, France
Locations (12):
- France (12):
  - Institut de Cancérologie de l'Ouest/Paul Papin, Angers
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de l'Ouest/Rene Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - INSTITUT DE CANCEROLOGIE Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut de Cancerologie de Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vanacker H, Treilleux I, Schiffler C, Bieche I, Campone M, Patsouris A, Arnedos M, Cottu PH, Jacquin JP, Dalenc F, Pinton A, Servant N, Attignon V, Rouleau E, Morel A, Legrand F, Jimenez M, Andre F, Bachelot T. p4EBP1 staining predicts outcome in ER-positive endocrine-resistant metastatic breast cancer patients treated with everolimus and exemestane. Br J Cancer. 2024 Mar;130(4):613-619. doi: 10.1038/s41416-023-02549-8. Epub 2024 Jan 5. PMID 38182687

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT02444390/SAP_000.pdf